CLINICAL TRIAL: NCT04302532
Title: Combined Coenzyme Q10 and Clomiphene Citrate for Ovulation Induction in Clomiphene-citrate-resistant Polycystic Ovary Syndrome
Brief Title: Coenzyme q 10 and Fertility Outcome in Women With Clomiphene Resistant PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karachi Medical and Dental College (Other)
Responsible Party: Principal Investigator, samia husain, clinical investigator, Karachi Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Coenzyme q10
Keywords: ovulation induction; coenzyme q10; pregnancy rate
MeSH Terms: interventions — coenzyme Q10; Clomiphene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clomiphene (Active Comparator): clomiphene citrate 150 mg once a day for 5 days
  Interventions: Drug: clomiphene citrate
- clomiphene and coenzyme q10 (Experimental): clomiphene citrate 150 mg once a day for 5 days and coenzyme q 10 120 mg each day
  Interventions: Drug: Coenzyme Q10; Drug: clomiphene citrate

INTERVENTIONS:
Drug: Coenzyme Q10 — antioxidant used to decrease oxidative stress and improve fertility prospects
  Other Names: celeron sr
  Arms: clomiphene and coenzyme q10
Drug: clomiphene citrate — ovulation induction drug
  Other Names: clomid

SUMMARY:
The study evaluates the effect of coenzyme q 10 on ovulation and subsequent pregnancy in women with polycystic ovarian syndrome. Half of the participants will receive coq10 and ovulation induction with clomiphene and other half would receive a placebo with clomiphene.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of polycystic ovarian syndrome PCOS based on the revised 2003 consensus on diagnostic criteria and long-term health risks related to PCOS (2003).
* All women were previously treated with 100 mg of CC daily for 5 days per cycle, for two to three cycles with persistent anovulation or ovulate with very thin endometrium <5 mm at the time of hCG administration

Exclusion Criteria:

* Non-consenting.
* known autoimmune disorders
* prior treatment of endometriosis or surgery to reproductive tract
* prior history of pelvic inflammatory disease
* those with tubal factors and uterine factors as assessed on history and confirmed by normal hysterosalpingogram.
* Thyroid disorder as assessed by history examination and TSH level
* Patients with raised FSH

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 149 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
number of ovulating women | 1-2 months
  transvaginal ultrasound as the disappearance of the leading follicle, presence of follicular fluid in the Douglas pouch and midluteal progesterone >5 pg/ml.
number of pregnancies | 1-2 months
  ultrasound visualization of gestational sac with pulsating fetal pole

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Izhar, Study Director — Aziz Medical Center
Locations (1):
- Aziz medical center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No